CLINICAL TRIAL: NCT06107348
Title: COVID-19 Post-Vaccination Observation on Immune Exhaustion
Brief Title: COVID-19 Post-Vaccination Observation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yang I. Pachankis, PhD (Individual)
Responsible Party: Sponsor-Investigator, Yang I. Pachankis, PhD, PI, Pachankis, Yang I., M.D.
Organization: Pachankis, Yang I., M.D. (Individual)
Other Study IDs: SARS-Immune-00
Record Dates: First submitted 2023-10-26; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Immune System Diseases; COVID-19 Vaccine Adverse Reaction; Immune System Disorder
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immune Disorder

SUMMARY:
The study started after the second COVID-19 vaccination of the participant with blood spots appearing on the skin with severe arthritis. The study continued to the third-dose full vaccination of the participant with the recombined COVID-19 vaccination and afterwards. The study completed until intervention.

ELIGIBILITY:
All COVID-19 vaccinated are eligible for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is currently focused on Asians.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-12-24 (Estimated)

PRIMARY OUTCOMES:
Chemiluminescent Immunoassay for Human Immunodeficiency Virus | 7 months
Carcinoembryonic Antigen | 7 months
Alpha Fetoprotein | 7 months
Carbohydrate Antigen 19-9 | 7 months
Mucin-16 | 7 months
Cancer Antigen 15-3 | 7 months
Prostate-Specific Antigen | 7 months
Leukocytes | 7 months
Leukocyte Percentage | 7 months
Cholesterol | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Residential Address, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: The data will be available upon completion and will be kept for as long as the repository is available.

REFERENCES:
- [Background] Pachankis YI. Questions of COVID-19: Institutional Derogations of Global Health. Lambert Academic Publishing. 2023. ISBN: 978-6206153849.
- Available data/document: Individual Participant Data Set: 10.17605/OSF.IO/2MGJK — http://doi.org/10.17605/OSF.IO/2MGJK